CLINICAL TRIAL: NCT04822623
Title: Computer Aided Imaging Evaluation of Central Nervous System Autoimmune Diseases
Brief Title: Imaging Evaluation of Central Nervous Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020SDUCRCC019
Record Dates: First submitted 2021-03-11; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-07

CONDITIONS: MS (Multiple Sclerosis); NMO Spectrum Disorder
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MS
  Interventions: Diagnostic Test: MRI
- NMOSD
  Interventions: Diagnostic Test: MRI
- Control
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI examination

SUMMARY:
Multiple sclerosis (MS) is the most common demyelinating disease of the central nervous system and the most common cause of non traumatic disability in young and middle-aged people. Neuromyelitis optica spectrum disease (nmosd) is an independent disease different from Ms. the pathogenesis and the mode of brain and spinal cord injury are different from MS, and the prognosis and optimal treatment are different. It is difficult to distinguish the two diseases in the early stage. Early diagnosis and treatment of the two diseases can greatly improve the quality of life of patients. Therefore, it is an urgent problem to clarify the difference between MS and nmosd injury patterns and to find sensitive imaging markers for early clinical intervention. With the continuous progress of computer aided diagnosis (CAD), it is more and more widely used in medicine, which is expected to help solve the above problems.

The purpose of this study is to create a neuroimmune disease evaluation database based on image data. By combining brain and spinal cord imaging, and based on Zhang quantum space learning computer-aided technology, we can achieve accurate segmentation of MS and nmosd brain and spinal cord lesions, analyze the evolution characteristics of the disease at different time points, and screen the imaging indexes related to clinical scores combined with clinical and laboratory indexes Objective: to determine the different prognosis and its influencing factors at the clinical, imaging and molecular levels, and establish the model for predicting disease progression and prognosis, so as to provide the basis for early identification and assistance in guiding treatment and judging prognosis.

Clinical information was collected: age, gender, course of disease, MMSE, EDSS disability score, nine hole test, 25 foot walking test. Assess the patient's information processing ability. Blood samples were collected. Imaging examination was performed. The patients were followed up regularly.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old;
2. Nmosd was diagnosed according to wingerchuk standard revised in 2015, MS was diagnosed according to McDonald standard revised in 2017, and 100 normal people were diagnosed;
3. In the acute stage, within 1 month of the onset or stable stage, there was no GD enhanced lesion on MRI, and EDSS score had no significant change within 6 months, which was more than 1 month from the last attack;
4. MRI examination was complete: baseline, 6 months, 1 year, 2 years;
5. Sign informed consent.

Exclusion Criteria:

1. The course of disease was more than 30 years;
2. History of brain injury or spinal cord injury;
3. History of central nervous system infection or immunodeficiency syndrome;
4. HBV, HCV patients, syphilis, HIV-1, HIV-2 patients;
5. Suffering from mental illness;
6. Pregnant and lactating women or patients planning to conceive within one year;
7. Unable to cooperate to complete the follow-up due to geographical or other reasons;
8. Patients also participated in other randomized controlled trials.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients in MS group and nmosd group were recruited from the Department of Neurology (outpatient and inpatient); the volunteers in control group were recruited through subject recruitment advertisement.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Results of MRI data analysis | 2021-03-01-2022-06-30
  The baseline data of MS, nmosd and normal group were complete, and the number of cases completed follow-up according to the requirements reached the expected requirements (100 cases each), and met the statistical standards.

IPD SHARING:
Plan to Share IPD: No